CLINICAL TRIAL: NCT00476372
Title: Cognitive Impairment in Parkinson's Disease Categorised in Accordance to Motor Symptoms -the Relation Between Cognitive Deficits and Comorbid Psychiatric Disorders, Medication, and Age at Disease Onset
Brief Title: Cognitive Impairment in Parkinson's Disease Categorised in Accordance to Motor Symptoms
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: UAarhus
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease
Keywords: neuropsychology; cognitive impairment; motor disorder; parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Motor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parkinson's disease: Pt with parkinsons disease

SUMMARY:
Background: Approximately 40% of patients with Parkinson's disease (PD) have cognitive impairments. There is a lack of consensus as to the extent to which psychiatric symptoms, depression, age at disease onset, disease duration, and medication is related to the type and severity of cognitive impairment. This discrepancy can in part be caused by the lack of distinction between patients with different motor symptoms and disease severity.

Objective: To identify the extent to which psychiatric symptoms, depression, age at disease onset, disease duration, and medication is related to the severity and type of cognitive dysfunction in patients with idiopathic PD categorized according to motor symptoms and disease severity.

Methods: the population of patients with PD in the old county of Aarhus is described on the background of medical records, and stratified in accordance to age, sex and cardinal symptoms. Through proportional allocation a sample of a minimum of 50 patients with PD is drawn from the population. The patients and 30 healthy matched controls will undergo comprehensive neuropsychological assessment including tests of language, memory, executive function, and visuospatial function. Furthermore, all participants will be screened for depression (Geriatric Depression Scale) and psychiatric symptoms (Neuropsychiatric Inventory and Symptom Checklist). The patients will be categorized in accordance with their motor symptoms via cluster analysis for the purpose of analyzing the effect of psychiatric symptoms, depression, and age of disease onset, disease duration, and medication on cognition.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's in accordance to UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria,
* Born and raised in Denmark ,
* >50 years

Exclusion Criteria:

* Cerebrovascular disease,
* Dementia not caused by Parkinson's Disease,
* Metabolism anomaly,
* Abuse of drugs, medication or alcohol,
* History of head injuries,
* Severe psychiatric disorder, excluding depression,
* Resident outside the region of Aarhus h) DBS -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 77 patients with PD and 30 healthy control participants
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
cognitive measures | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Karen Østergaard, neurologist, Study Chair — Aarhus University Hospital; Lars Larsen, MSc, PhD, Associate Professor, Study Chair — The Institute of Psychology
Locations (1):
- Aarhus Universitetshospital, Aarhus, Denmark